CLINICAL TRIAL: NCT06064435
Title: Safety and Efficacy of Endovascular Coiling Using Target Tetra® Coils for Small Intracranial Aneurysm: Prospective, Open-label, Single Arm, Single Center Study
Brief Title: Endovascular Coiling Using Target Tetra® Coils for Small Intracranial Aneurysm
Status: Not yet recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2023-0053
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Intracranial Aneurysm
Keywords: Small intralcranial aneurysm; Target Tetra Coils
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tetral Coil Group: Intracranial Aneurysm patients who treated with Target Tetra® coils (70% or more of packing density)

SUMMARY:
The goal of this study was to verify the safety and effectiveness of Target Tetra® Detachable Coil in the endovascular embolization treatment of small intracranial aneurysm (≤5mm).

DETAILED DESCRIPTION:
The study is a Prospective Single-arm Single-center Registry that aims to assess the safety and efficacy of the Target Tetra Coils in the endovascular treatment of small intracranial aneurysms (≤5mm). The study is not designed as intervention or treatment study. The investigators will enroll up to 100 participants at the single center.

* Enrollment of patients: The following process is carried out for patients who have consented to participate in the study among non-ruptured or ruptured cerebral aneurysm patients selected based on the inclusion and exclusion criteria.

  * Before the procedure, the following items are verified:

    * Informed consent form
    * Demographic information
    * Past medical history and family history
    * Vital signs
    * Electrocardiogram (ECG) results (results from within the previous 12 weeks before the screening visit can be used)
    * Laboratory test results (results from within the previous 12 weeks before the screening visit can be used): WBC, RBC, Hb, Hct, platelet count, PT INR, aPTT, cholesterol, ALP, AST, ALT, albumin, total bilirubin, total protein, BUN, creatinine, eGFR*, Urine-HCG†, FBS, triglycerides, LDL, PRU (VerifyNow test), and ARU (VerifyNow test) *eGFR = (140 - age) x (weight/72) x Creatinine

      * Pregnancy test (if applicable)
    * Imaging findings (results from within the previous 1 year before the screening visit can be used)
    * Adverse events
    * Concomitant medications/therapies
    * Pre-procedure modified Rankin Scale (mRS) assessment

      ③ Following the established method, coil embolization is performed under general anesthesia, and mechanical or technical failures of the Target Tetra® Detachable Coil occurring during the treatment are investigated.
    * Failure to advance or insert
    * Stretch
    * Disconnection
    * Detachment failure
    * Material deformation
    * Difficult to remove
    * Peeled or delaminated device
    * Premature detachment ④ During the procedure and within 30 days post-procedure, neurological and non-neurological complications are investigated.
    * Neurological complications

      -Any cause of death
      * Any intracranial thromboembolism (asymptomatic or symptomatic)
      * Any intracranial hemorrhage including aneurysm perforation
      * Any intracranial vessel injury
      * Miscellaneous: any ocular hemorrhage
    * Non-neurological complications

      -Puncture site complication requiring any intervention

      -Pseudoaneurysm

      -Arteriovenous (AV) fistula

      -Hematoma requiring transfusion

      -Retroperitoneal hemorrhage

      -Arterial dissection
      * Thromboembolism including limb ischemia
      * Miscellaneous: infection, vessel rupture/perforation
      * Complications related to general anesthesia

        * After the procedure, the occlusion rate of cerebral aneurysms (modified Raymond Scale; complete occlusion, neck remnant, sac remnant) and packing density are evaluated.
    * Modified Raymond Scale
    * Packing Density Packing Density = Volume of coils placed in the aneurysm / Volume of the aneurysm measured on a 3D workstation (%) The above process is conducted through the open-source Angiosuite application.

      ⑥ Characteristics of cerebral aneurysms in patients who have been treated with Target Tetra® Detachable Coils in over 70% of the total packing density are identified.

      ⑦ Clinical outcomes (mRS) are evaluated at 1 month, 6 months, 12 months of follow-up.

<Modified Rankin Scale score>

⑧ At 6 months, 12 months, the occlusion rate of cerebral aneurysms (Modified Raymond Scale) and recurrence are assessed by at least two neurosurgery specialists using 3T-MR angiography or cerebral angiography.

⑨ Patients who have not been treated with Target Tetra® Detachable Coils in over 70% of the total packing density are excluded from the analysis.

The independent Study Monitoring will be regularly proceed and processed on the basis of the permission of instituitional review board.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 to 80 years
2. Patients with intracranial aneurysms suitable for endovascular embolization therapy with a maximum diameter of 5mm or less
3. Including both ruptured and unruptured intracranial aneurysms
4. Patients for whom the use of Target Tetra® coil is expected in endovascular coil embolization therapy
5. Patients who have undergone balloon-assisted coiling or adjunctive stent placement during coil embolization
6. Subjects who have received an explanation of the clinical study and provided written consent to participate in the study

Exclusion Criteria:

1. Age below 18 or above 81 years
2. Infectious, dissecting, traumatic, or mycotic aneurysms
3. Patients who have undergone surgical or endovascular treatment for the target intracranial aneurysm
4. Patients in whom vascular access to the target intracranial aneurysm is not possible due to conditions such as moyamoya disease, dural arteriovenous malformation, significant atherosclerotic stenosis, or severe vessel tortuosity
5. Patients with ruptured intracranial aneurysms classified as Hunt and Hess grade 5 (deep coma)
6. Patients with hypersensitivity reactions to the materials used in the coils, such as platinum, tungsten, nickel, or stainless steel
7. Patients with serious adverse reactions to contrast agents
8. Patients who are unable to complete planned follow-up observations due to expected short-term survival or comorbidities
9. Female patients who are pregnant (positive pregnancy test) or planning pregnancy within 12 months after coil placement, or breastfeeding
10. Patients with significant renal dysfunction or uncorrected coagulation disorders

Ages: 19 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with small-sized intracranial aneurysms measuring 5mm or less require endovascular coil embolization treatment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Anerysm Occlusion Grade : Procedure day Occlusion Grade | Procedure day
Anerysm Occlusion Grade : 6 month Occlusion Grade | 6 months(±30 days) from procedure date
Anerysm Occlusion Grade : 12 month Occulsion Grade | 12 months(±30 days) from procedure date
Aneurysm Packing Density : Packing Density | Procedure day

SECONDARY OUTCOMES:
Neurological complications | Procedure, 1 month from procedure date
  Neurological complications related to the use of the device during the procedure
Non-neurological complications | Procedure, 1 month from procedure date
  Non-neurological complications related to the use of the device during the procedure
Device-related events | procedure date
  Device-related events during the procedure (malfunction, stretching, early detachment, etc.)
Clinical outcomes | Procedure, 1 month, 6 months, 12 months from procedure date
  Clinical outcomes observed during the follow-up perio
Incidence of recurrence and retreatment | Procedure, 6 months, 12 months from procedure date
  Incidence of recurrence and retreatment during the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Keunyoung PARK, M.D.PhD., Principal Investigator — Department of Neurosurgery, Yonsei University College of Medicine, Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No